CLINICAL TRIAL: NCT04530877
Title: Comparative Effectiveness of Exclusive Enteral Nutrition and Infliximab in Chinese Children With Active Crohn's Disease
Brief Title: Exclusive Enteral Nutrition vs. Infliximab in Chinese CD Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: no funding
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Ying HUANG, Director, Children's Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: twj01
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2022-08-09 (Actual); Status verified 2022-08

CONDITIONS: Crohn's Disease; Exclusive Enteral Nutrition; Infliximab; Mucosal Healing
MeSH Terms: conditions — Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exclusive enteral nutrition (Experimental): the administration of a liquid formula diet with the exclusion of all other regular food for 8 weeks， the volume was determined according to the energy needs of the patient. All patients received high energy intakes (>110%-120% of the average requirement).
  Interventions: Dietary Supplement: Exclusive Enteral Nutrition
- Infliximab (Active Comparator): the participants with active CD accept anti-TNF therapy (Infliximab) at 0week, 2week, 6week, 14week. Infliximab, a monoclonal antibody-targeting tumor necrosis factor (TNF), is one of the primary treatment strategies for active pediatric CD
  Interventions: Biological: Infliximab

INTERVENTIONS:
Biological: Infliximab — Infliximab, a monoclonal antibody-targeting tumor necrosis factor (TNF), is one of the primary treatment strategies for active pediatric CD
  Arms: Infliximab
Dietary Supplement: Exclusive Enteral Nutrition — the administration of a liquid formula diet with the exclusion of all other regular food for 6-8 weeks， the volume was determined according to the energy needs of the patient. All patients received high energy intakes (>110%-120% of the average requirement).
  Arms: Exclusive enteral nutrition

SUMMARY:
prospectively compared Exclusive Enteral Nutrition with Infliximab in the clinical outcomes, mucosal healing, nutrition improvements, adverse effects and gastrointestinal microbiota changes on Chinese Children With active Crohn's Disease

ELIGIBILITY:
Inclusion Criteria:

patients:

1. Pediatric active Crohn's disease ( CD) patients who were newly diagnosed at the Children's Hospital of Fudan University from October 2020 to Sep 2022，CD was diagnosed according to the Porto criteria and based on a combination of history, physical and laboratory examination, endoscopy with histology, and imaging of the small bowel (capsule endoscopy or magnetic resonance imaging or enhanced computerized tomography).
2. SES-CD>4 and PCDAI >10 at initial
3. For the patients whose fecal will be analyzed shouldn't take antibiotics or probiotics within the 1.5 months prior to the study and during the treatment.

healthy controls:

1. free medical history
2. had not taken antibiotics or probiotics within the 1.5 months prior to donate their fecal

Exclusion Criteria:

1. patients who had gene mutation or combined with other intestinal diseases such as tuberculosis or EB infection
2. for patients in the EEN group who could not finish the daily prescribed volume of formula for any reason; for the patients in the IFX group who could not finish the first 4 times IFX injection for any reason.
3. patients who were administered EEN, corticosteroids, immunosuppressive drugs, or biological agents prior to the study;
4. patients who could not attend consecutive follow-up sessions;

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
the number of patients who reach mucosal healing at the end of treatment in Exclusive enteral nutrition group | at the end of 8 week of treatment.
  the mucosal healing was defined as Simple Endoscopic Score for CD （SES-CD ）≤4 at the end of treatment . For the SES-CD, the intestine is divided into 5 anatomic segments under the endoscopic vision: rectum, left side of the colon segment, transverse colon, right side of the colon segment, and ileum. Items of interest include ulcer size, estimates of the ulcerated and affected surface, and the presence of luminal narrowing. The SES-CD score is calculated by combining scores of individual segments. Overall SES-CD scores are classified into 4 disease categories: none, 0 to 2; mild 2 to 4; moderate 5 to 15; and severe>16.
the number of patients who reach mucosal healing at the end of treatment in Infliximab group | at the end of 14 week of treatment.
  the mucosal healing was defined as Simple Endoscopic Score for CD （SES-CD ）≤4 at the end of treatment . For the SES-CD, the intestine is divided into 5 anatomic segments under the endoscopic vision: rectum, left side of the colon segment, transverse colon, right side of the colon segment, and ileum. Items of interest include ulcer size, estimates of the ulcerated and affected surface, and the presence of luminal narrowing. The SES-CD score is calculated by combining scores of individual segments. Overall SES-CD scores are classified into 4 disease categories: none, 0 to 2; mild 2 to 4; moderate 5 to 15; and severe>16.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Huang, Dr, Study Chair — Department of Gastroenterology, Pediatric Inflammatory Bowel Disease Research Center, Children's Hospital of Fudan University